CLINICAL TRIAL: NCT06757881
Title: A Phase 1 Study of IL1RAP-targeting Chimeric Antigen Receptor T Cells in the Treatment of Relapsed/Refractory Hepatocellular Carcinoma
Brief Title: IL1RAP-targeting Chimeric Antigen Receptor T Cells in the Treatment of Relapsed/Refractory Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-272(2)
Record Dates: First submitted 2024-12-20; First posted 2025-01-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: HCC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gene modified anti-IL1RAP Chimeric Antigen Receptor T Cells (Experimental)
  Interventions: Biological: Gene modified anti-IL1RAP Chimeric Antigen Receptor T Cells :1.0×10^8(First dose group); Biological: Gene modified anti-IL1RAP Chimeric Antigen Receptor T Cells :2.5×10^8(Second dose group); Biological: Gene modified anti-IL1RAP Chimeric Antigen Receptor T Cells :5.0×10^8（Third dose group）

INTERVENTIONS:
Biological: Gene modified anti-IL1RAP Chimeric Antigen Receptor T Cells :1.0×10^8(First dose group) — Different dose groups
Biological: Gene modified anti-IL1RAP Chimeric Antigen Receptor T Cells :2.5×10^8(Second dose group) — Different dose groups
Biological: Gene modified anti-IL1RAP Chimeric Antigen Receptor T Cells :5.0×10^8（Third dose group） — Different dose groups

SUMMARY:
A Phase 1 Study of IL1RAP-targeting Chimeric Antigen Receptor T cells in the Treatment of Relapsed/Refractory Hepatocellular Carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years old, male or female;
2. Patients with advanced hepatocellular carcinoma who are confirmed by histopathology and/or cytology to be ineligible for surgery and local radical therapy and who have developed tumor progression or toxicity intolerance following at least one standardized systemic therapy (including molecularly targeted agents and immune checkpoint inhibitors) or interventional therapy
3. Liver cancer subjects with stage II or III of China Liver Cancer Staging (CNLC) as defined by Barcelona Clinic Liver Cancer (BCLC) B/C level or the Code of Practice for Primary Liver Cancer Diagnosis and Treatment (2022 edition);
4. Expected survival ≥3 months
5. Before the start of the research related procedures, after explaining the research content, voluntarily participate and be able to sign the informed consent; Agree to and have the ability to follow study visits, imaging tests, laboratory tests, and other research procedures in the study plan;
6. Good compliance, willing and able to follow all research procedures, and cooperate with observation and follow-up.

Exclusion Criteria:

1. Have had other uncured malignancies within the past 5 years or at the same time, except for in situ cancers considered clinically curable, such as cervical carcinoma in situ and basal cell carcinoma of the skin
2. Central nervous system metastases and clinically significant central nervous system diseases
3. Pregnant or lactating women;
4. The investigator believes that the subjects have any circumstances that make them unfit to participate in this clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limited Toxicity | Within 28 days after the cell infusion
Number of participants with treatment associated adverse events (AE) and serious adverse events (SAE) according to CTCAE v5.0 | From the start of PBMC collection until subject withdrawal or 12 months after cell infusion, participants who withdraw without cell infusion will be only collected for AEs within 28 days after the study-related procedure or other treatment begins
Number of participants with cytokine release syndrome (CRS) and immune effector cell-associated neurotoxicity syndrome (ICANS) | From the start of PBMC collection until subject withdrawal or 12 months after cell infusion, participants who withdraw without cell infusion will be only collected for AEs within 28 days after the study-related procedure or other treatment begins
Number of participants with treatment associated changes in clinically significant laboratory safety test values | From the start of PBMC collection until subject withdrawal or 12 months after cell infusion, participants who withdraw without cell infusion will be only collected for AEs within 28 days after the study-related procedure or other treatment begins

SECONDARY OUTCOMES:
Curative effect evaluation | 3 months after cell infusion
  3-month objective response rate (ORR); 、
Disease control rate (DCR) | 3 months, 6 months, 1 year, 2years after cell infusion
Changes of serum IL1RAP level | 3 months, 6 months, 1 year, 2years after cell infusion
Changes of copy number and absolute value of CAR-T cells targeting IL1RAP in peripheral blood | 3 months, 6 months, 1 year, 2years after cell infusion
Progression-free survival (PFS) | 3 months, 6 months, 1 year, 2years after cell infusion
Median PFS | 3 months, 6 months, 1 year, 2years after cell infusion
Time to remission (TTR) | 3 months, 6 months, 1 year, 2years after cell infusion
Duration of response after administration (DOR) | 3 months, 6 months, 1 year, 2years after cell infusion
Survival time: Median overall survival (mOS) | 6 months, 1 year, 2years after cell infusion
OS rate | 6 months, 1 year, 2years after cell infusion
PFS rate | 3 months, 6 months, 1 year, 2years after cell infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No